CLINICAL TRIAL: NCT01781130
Title: Effect of Steroid Injection Which is Added to Percutaneous Trigger Finger Release: a Double-blinded Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Min Jong Park, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-11-112-002
Record Dates: First submitted 2013-01-15; First posted 2013-01-31 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Trigger Finger
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Steroids

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Percutaneous release alone (Placebo Comparator): The patients who perform percutaneous release of trigger finger only
- Percutaneous release + Steroid injection (Experimental): Steroid local injection after percutaneous release of trigger finger
  Interventions: Procedure: Steroid injection

INTERVENTIONS:
Procedure: Steroid injection
  Arms: Percutaneous release + Steroid injection

SUMMARY:
Background

Present treatment strategies for trigger finger when conservative management including steroid injection was failed include percutaneous or open A1 pulley release, but some people showed prolonged swelling and delay of complete healing.

We aimed to test the hypothesis that an improved outcome can be achieved by employing steroid injection simultaneously with percutaneous release compared with conventional percutaneous release alone

Methods

We designed a double-blind, randomized controlled trial.

Inclusion criteria is the patient who has symptom of trigger finger warranted surgical release after sufficient time of conservative treatment.

Exclusion criteria are as follow: 1) multiple fingers at presentation; 2) Rheumatoid arthritis patients; 3) Pregnant or lactating patients; 4) Younger than 18 years old; 5) Previous surgery history of finger 6); the patients who got steroid injection more than 4 time previously; 7) coagulation abnormality including usage of anti-thrombotic agent.

After power analysis by a statistician, total 40 patients would be required for each group (percutaneous alone group versus percutaneous alone + steroid injection group).

The surgery will be performed by outpatients clinic basis with local injection. Additional steroid injection will be given to half of patients after allocation with randomized selection by permutaed block randomization.

Primary outcome measure is mean fall in pain visual analogue scale (pVAS) and secondary outcome will be proportion of patients with good response (defined as "Perfect" or "much better" as reported by patients).

Follow-up will be conducted 3 weeks and 3 month after index procedure

ELIGIBILITY:
Inclusion Criteria:

* Trigger finger patients who require surgical intervention due to failuer of sufficient time of conservative treatment

Exclusion Criteria:

* Age under 18 years old
* Rheumatoid arthritis patients
* Patients who got steroid injection more than 4 times previously
* Multiple finger affected at presentation
* Previous surgery history
* Any recent trauma history of affected hand

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
pain VAS | 3 month after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Patel MR, Moradia VJ. Percutaneous release of trigger digit with and without cortisone injection. J Hand Surg Am. 1997 Jan;22(1):150-5. doi: 10.1016/S0363-5023(05)80196-0. PMID 9018629